CLINICAL TRIAL: NCT01656239
Title: A Randomised, Double-Blind, Placebo-Controlled, Parallel Group, Dose Range Finding Study To Determine The Efficacy And Safety Of Fedovapagon In Men With Nocturia
Brief Title: Dose Range Finding Study of Fedovapagon in Men With Nocturia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vantia Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 483-009
Record Dates: First submitted 2012-07-31; First posted 2012-08-02 (Estimated); Last update posted 2014-06-20 (Estimated); Status verified 2014-06

CONDITIONS: Nocturia
Keywords: VA106483, fedovapagon, Nocturia, males, nocturnal voids, anti-diuretic
MeSH Terms: conditions — Nocturia | interventions — Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- fedovapagon 1 mg (Experimental): Once daily oral dose of 1 mg fedovapagon for 12 weeks
  Interventions: Drug: fedovapagon 1 mg
- fedovapagon 2 mg (Experimental): Once daily oral dose of 2 mg fedovapagon for 12 weeks
  Interventions: Drug: fedovapagon 2 mg
- fedovapagon 4 mg (Experimental): Once daily oral dose of 4 mg fedovapagon for 12 weeks
  Interventions: Drug: fedovapagon 4 mg
- sugar pill (Placebo Comparator): Once daily oral dose of placebo for 12 weeks
  Interventions: Drug: Placebo ( sugar pill)

INTERVENTIONS:
Drug: fedovapagon 1 mg
  Arms: fedovapagon 1 mg
Drug: fedovapagon 2 mg
  Arms: fedovapagon 2 mg
Drug: fedovapagon 4 mg
  Arms: fedovapagon 4 mg
Drug: Placebo ( sugar pill)
  Arms: sugar pill

SUMMARY:
The purpose of this study is to determine the dose level(s) of fedovapagon which result in a decrease in the mean nocturnal void frequency.

DETAILED DESCRIPTION:
Fedovapagon is a selective vasopressin V2 receptor (V2 receptor) agonist that is being developed for the treatment of Nocturia.

The antidiuretic effect of V2 receptor stimulation in the kidneys is well established through the use of the peptide agonist, desmopressin, which shows clinical benefit in diabetes insipidus, primary nocturnal enuresis and Nocturia.

Nocturia, defined as the complaint that the individual has to wake at night one or more times to void, is a common complaint and shows an age-dependent increase in both prevalence and severity (number of Nocturnal Voids). It is the most bothersome symptom of benign prostatic hypertrophy (BPH) and has been linked to an age-dependent loss in circadian release of endogenous nocturnal vasopressin and consequent over production of urine at night (Nocturnal Polyuria).

The purpose of this Phase IIb study is to determine the efficacy of different doses of fedovapagon in reducing the number of times subjects with Nocturia void during the night together with other parameters including increasing the time between going to bed and waking to first void. By establishing the effective doses of fedovapagon on these clinical endpoints, the data from this study will determine the most appropriate dose(s) of fedovapagon for the treatment of Nocturia to be taken forward into further studies.

ELIGIBILITY:
Inclusion Criteria:

* Males aged 55 or over
* History and/ or symptoms of Nocturia (2 - 5 voids per night)
* Generally well (concomitant illness / conditions well controlled)
* Serum sodium, potassium, chloride and bicarbonate within normal limits
* No clinically significant abnormalities in other laboratory parameters, urinalysis, electrocardiogram (ECG) or physical examination
* Prostate specific antigen (PSA) within the normal range or not considered clinically significant
* Ability to comply with the requirements of the study
* Written informed consent.

Exclusion Criteria:

-

Min Age: 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 358 (Actual)
Dates: Start 2012-08; Primary Completion 2013-08 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Change in the mean nocturnal urine voids | 12 weeks

SECONDARY OUTCOMES:
Change in the mean nocturnal urine voids | 4 weeks
Change in the mean time to first nocturnal void | 4 weeks
Change in the mean time to first nocturnal void | 12 weeks
Change in Nocturia-related quality of life (N-QOL) | 4 weeks
Change in Nocturia-related quality of life (N-QOL) | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hilary McElwaine-Johnn, BSc, ASM, MBBS, MRCP, MFPM, Study Director — Vantia Ltd
Locations (56):
- United States (56):
  - Vantia Investigative Center, Birmingham, Alabama
  - Vantia Investigative Center, Huntsville, Alabama
  - Vantia Investigative Center, Mobile, Alabama
  - Vantia Investigative Center, Glendale, Arizona
  - Vantia Investigative Center, Tucson, Arizona
  - Vantia Investigative Center, Anaheim, California
  - Vantia Investigative Center, Long Beach, California
  - Vantia Investigative Center, San Diego, California
  - Vantia Investigative Center, Denver, Colorado
  - Vantia Investigative Center, Englewood, Colorado
  - Vantia Investigative Center, Milford, Connecticut
  - Vantia Investigative Center, Aventura, Florida
  - Vantia Investigative Center, Clearwater, Florida
  - Vantia Investigative Center, Daytona Beach, Florida
  - Vantia Investigative Center, DeLand, Florida
  - Vantia Investigative Center, Naples, Florida
  - Vantia Investigative Center, Ocala, Florida
  - Vantia Investigative Center, St. Petersburg, Florida
  - Vantia Investigative Center, Tampa, Florida
  - Vantia Investigative Center, Coeur d'Alene, Idaho
  - Vantia Investigative Center, Meridian, Idaho
  - Vantia Investigative Center, Chicago, Illinois
  - Vantia Investigative Center, Evansville, Indiana
  - Vantia Investigative Center, Jeffersonville, Indiana
  - Vantia Investigative Center, Paducah, Kentucky
  - Vantia Investigative Center, Metairie, Louisiana
  - Vantia Investigative Center, Greenbelt, Maryland
  - Vantia Investigative Center, Rochester, Michigan
  - Vantia Investigative Center, Edina, Minnesota
  - Vantia Investigative Center, Omaha, Nebraska
  - Vantia Investigative Center, Brick, New Jersey
  - Vantia Investigative Center, Englewood, New Jersey
  - Vantia Investigative Center, Lawrenceville, New Jersey
  - Vantia Investigative Center, Albuquerque, New Mexico
  - Vantia Investigative Center, Brooklyn, New York
  - Vantia Investigative Center, Endwell, New York
  - Vantia Investigative Center, Garden City, New York
  - Vantia Investigative Center, New York, New York
  - Vantia Investigative Center, Poughkeepsie, New York
  - Vantia Investigative Center, Concord, North Carolina
  - Vantia Investigative Center, Raleigh, North Carolina
  - Vantia Investigative Center, Winston-Salem, North Carolina
  - Vantia Investigative Center, Cincinnati, Ohio
  - Vantia Investigative Center, Bethany, Oklahoma
  - Vantia Investigative Center, Bala-Cynwyd, Pennsylvania
  - Vantia Investigative Center, Warwick, Rhode Island
  - Vantia Investigative Center, Mytrle Beach, South Carolina
  - Vantia Investigative Center, Dakota Dunes, South Dakota
  - Vantia Investigative Center, Nashville, Tennessee
  - Vantia Investigative Center, Dallas, Texas
  - Vantia Investigative Center, Fort Worth, Texas
  - Vantia Investigative Center, San Antonio, Texas
  - Vantia Investigative Center, Richmond, Virginia
  - Vantia Investigative Center, Virginia Beach, Virginia
  - Vantia Investigative Center, Burien, Washington
  - Vantia Investigative Center, Middleton, Wisconsin